CLINICAL TRIAL: NCT02032524
Title: An Open-label, Multicenter, Multinational Extension Study of the Long-term Safety and Pharmacokinetics of Repeated Biweekly Infusions of Avalglucosidase Alfa (neoGAA, GZ402666) in Patients With Pompe Disease
Brief Title: Avalglucosidase Alfa Extension Study
Acronym: NEO-EXT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS13769; U1111-1147-3439 (Other: UTN)
Record Dates: First submitted 2013-12-04; First posted 2014-01-10 (Estimated); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Glycogen Storage Disease Type II Pompe Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avalglucosidase Alfa (Experimental): administered intravenously every 2 weeks
  Interventions: Drug: Avalglucosidase Alfa

INTERVENTIONS:
Drug: Avalglucosidase Alfa — Pharmaceutical form: lyophilized powder reconstituted for infusion Route of administration: intravenous
  Other Names: GZ402666; neoGAA

SUMMARY:
Primary Objective:

Long-term safety and pharmacokinetics (PK) of avalglucosidase alfa

Secondary Objective:

Long-term effect of avalglucosidase alfa on pharmacodynamic variables

DETAILED DESCRIPTION:
The planned duration of the study for each participant was initially 6 years. Each participant continued with the study until the participant withdrew, the Investigator withdrew the participant, or the Sponsor terminated the study. An additional follow-up phase began after the participant has completed the 6-year study period, and lasted until avalglucosidase alfa was approved in the participant's country, except in the United Kingdom (UK), Germany and Denmark, where the duration of the additional follow-up phase was up to the approval in the country or limited to a maximum of 2 years, whichever occurred first (ie, for participants in the UK, Germany and Denmark, the total study duration per participant was 8 years at the maximum including the initial 6-year period and the additional 2-year follow-up).

ELIGIBILITY:
Inclusion criteria:

Participants with Pompe disease who previously completed an avalglucosidase study.

The participant and/or their parent/legal guardian is willing and able to provide signed informed consent, and the participant, if <18 years of age, was willing to provide assent if deemed able to do so.

The participant (and participant's legal guardian if participant is <18 years of age) must have had the ability to comply with the clinical protocol.

The participant, if female and of childbearing potential, had to have a negative pregnancy test [urine beta-human chorionic gonadotropin] at baseline.

Exclusion criteria:

The participant was concurrently participating in another clinical study using investigational treatment.

The participant, in the opinion of the Investigator, was unable to adhere to the requirements of the study.

The participant had clinically significant organic disease (with the exception of symptoms relating to Pompe disease), including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, precluded participation in the study or potentially decreases survival.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02-27 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (17):
- United States (8):
  - Investigational Site Number 840006, Phoenix, Arizona
  - Investigational Site Number 840010, Jacksonville, Florida
  - Investigational Site Number 840001, Kansas City, Kansas
  - Investigational Site Number 840008, St Louis, Missouri
  - Investigational Site Number 840002, Durham, North Carolina
  - Investigational Site Number 840011, Cincinnati, Ohio
  - Investigational Site Number 840009, Dallas, Texas
  - Investigational Site Number 840003, Fairfax, Virginia
- Investigational Site Number 056001, Leuven, Belgium
- Investigational Site Number 208001, København Ø, Denmark
- France (2):
  - Investigational Site Number 250003, Nice
  - Investigational Site Number 250002, Paris
- Germany (3):
  - Investigational Site Number 276003, Mainz
  - Investigational Site Number 276001, München
  - Investigational Site Number 276002, Münster
- Investigational Site Number 528001, Rotterdam, Netherlands
- Investigational Site Number 826003, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Dimachkie MM, Barohn RJ, Byrne B, Goker-Alpan O, Kishnani PS, Ladha S, Laforet P, Mengel KE, Pena LDM, Sacconi S, Straub V, Trivedi J, Van Damme P, van der Ploeg AT, Vissing J, Young P, Haack KA, Foster M, Gilbert JM, Miossec P, Vitse O, Zhou T, Schoser B; NEO-EXT investigators. Long-term Safety and Efficacy of Avalglucosidase Alfa in Patients With Late-Onset Pompe Disease. Neurology. 2022 Aug 1;99(5):e536-e548. doi: 10.1212/WNL.0000000000200746. PMID 35618441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 centers in 7 countries. A total of 21 participants completed the open-label study TDR12857 (NCT01898364). Of which, 19 participants were enrolled in this study. There was no screening period in this study.
Pre-assignment Details: Participants who completed the open-label TDR12857 study were part of this study. This was an open-label study. As prespecified, data were analyzed and presented combinedly for studies TDR12857 and LTS13769.
Groups:
- Group 1: Avalglucosidase Alfa 5 mg/kg: Participants who were treatment-naïve to alglucosidase alfa received avalglucosidase alfa 5 milligram per kilogram (mg/kg) intravenous (IV) infusion every other week (qow) for up to 454 weeks.
- Group 1: Avalglucosidase Alfa 10 mg/kg: Participants who were treatment-naïve to alglucosidase alfa received avalglucosidase alfa 10 mg/kg IV infusion qow for up to 432 weeks.
- Group 1: Avalglucosidase Alfa 20 mg/kg: Participants who were treatment-naïve to alglucosidase alfa received avalglucosidase alfa 20 mg/kg IV infusion qow for up to 421 weeks.
- Group 2: Avalglucosidase Alfa 5 mg/kg: Participants who were previously treated with alglucosidase alfa received avalglucosidase alfa 5 mg/kg IV infusion qow for up to 424 weeks.
- Group 2: Avalglucosidase Alfa 10 mg/kg: Participants who were previously treated with alglucosidase alfa received avalglucosidase alfa 10 mg/kg IV infusion qow for up to 450 weeks.
- Group 2: Avalglucosidase Alfa 20 mg/kg: Participants who were previously treated with alglucosidase alfa received avalglucosidase alfa 20 mg/kg IV infusion qow for up to 445 weeks.
Period: Period 1: TDR12857 Study
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Started | 4 | 3 | 3 | 4 | 4 | 6
Completed | 3 | 3 | 3 | 3 | 4 | 5
Not Completed | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Wishes To Withdraw | 0 | 0 | 0 | 1 | 0 | 1
Period: Period 2: LTS13769 Study
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Started (Enrolled and treated participants in LTS13769 study.) | 3 | 2 (Only eligible participants enrolled in LTS13769 study.) | 3 | 3 | 3 (Only eligible participants enrolled in LTS13769 study.) | 5
Completed | 3 | 1 | 2 | 3 | 2 | 4
Not Completed | 0 | 1 | 1 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Wishes To Withdraw | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis (FA) set included all participants who received at least 1 complete infusion of investigational medicinal product (IMP).
Groups:
- Group 1: Avalglucosidase Alfa 5 mg/kg: Participants who were treatment-naïve to alglucosidase alfa received avalglucosidase alfa 5 mg/kg IV infusion qow for up to 454 weeks.
- Total: Total of all reporting groups
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg | Total
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants] — Age at TDR12857 inform consent.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 3 | 3 | 2 | 3 | 4 | 5 | 20
    >=65 years | 1 | 0 | 1 | 1 | 0 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 2 | 1 | 2 | 12
  Male | 1 | 0 | 2 | 2 | 3 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 1 | 3 | 4 | 3 | 6 | 21
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Multiple | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), Infusion Associated Reactions (IARs) and Deaths
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An serious AE (SAE) is any untoward medical occurrence that results: death or life-threatening or inpatient hospitalization or prolongation of existing hospitalization or persistent or significant disability or congenital anomaly or medically important event. TEAEs are defined as AEs that develop or worsen during the on-treatment period (that is, from the time of first dose of IMP up to 4 weeks after the last administration of the IMP). Protocol-defined IARs were defined as AEs that occur during either the infusion or the post-infusion observation period (that is, up to 2 hours or longer following the infusion as per the Investigator's discretion) which were deemed to be related or possibly related to the IMP.
Time Frame: From first dose of IMP up to 4 weeks after the last treatment administration of the IMP, a maximum up to 458 weeks
Population: The safety analysis set included all participants who received at least 1 complete infusion of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
Participants
  Any TEAEs | 4 | 3 | 3 | 4 | 4 | 6
  TESAEs | 3 | 1 | 1 | 1 | 1 | 2
  Protocol-defined IARs | 2 | 0 | 2 | 2 | 0 | 1
  Any TEAE leading to death | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities
Description: Physical examination included, at a minimum, an assessment of the participant's general appearance; skin; head, eyes, ears, nose, and throat; examinations of lymph nodes, abdomen, extremities/joints, neurological and mental status; heart and respiratory auscultation; peripheral arterial pulse; and pupil, knee, achilles, and plantar reflexes.
Time Frame: From first dose of IMP up to 4 weeks after the last treatment administration of the IMP, a maximum up to 458 weeks
Population: The safety analysis set included all participants who received at least 1 complete infusion of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
Participants
  Achilles Reflexes | 0 | 0 | 0 | 0 | 0 | 1
  General Appearance | 0 | 0 | 0 | 0 | 0 | 1
  Knee Reflexes | 0 | 0 | 0 | 0 | 0 | 1
  Lymph Nodes | 0 | 0 | 0 | 0 | 0 | 1
  Neurological Status | 0 | 0 | 0 | 0 | 2 | 1

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities in Biochemistry
Description: Blood samples were collected to determine the clinical chemistry laboratory abnormalities.
Time Frame: From first dose of IMP up to 4 weeks after the last treatment administration of the IMP, a maximum up to 458 weeks
Population: The safety analysis set included all participants who received at least 1 complete infusion of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
Participants
  Glucose: <=3.9 millimoles per liter (mmol/L) and < lower limit of normal (LLN) | 2 | 2 | 2 | 1 | 2 | 1
  Glucose: >=11.1 mmol/L (unfasted); >=7 mmol/L (fasted) | 2 | 0 | 1 | 1 | 1 | 3
  Sodium: <=129 mmol/L | 0 | 0 | 0 | 1 | 0 | 1
  Sodium: >=160 mmol/L | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: <3 mmol/L | 0 | 0 | 0 | 1 | 1 | 0
  Potassium: >=5.5 mmol/L | 0 | 0 | 0 | 0 | 0 | 1
  Chloride: <80 mmol/L | 0 | 0 | 0 | 0 | 0 | 0
  Chloride: >115 mmol/L | 0 | 0 | 0 | 0 | 0 | 0
  Albumin: <=25 gram per liter (g/L) | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: >=150 micromoles/L (Adults) | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine: >=100% change from baseline | 0 | 0 | 0 | 0 | 0 | 2
  Creatinine: >=30% change from baseline | 0 | 0 | 0 | 1 | 0 | 2
  Urea Nitrogen: >=17 mmol/L | 0 | 0 | 1 | 0 | 0 | 0
  Aspartate Aminotransferase: >3 upper limit of normal (ULN) | 0 | 2 | 0 | 1 | 0 | 0
  Aspartate Aminotransferase: >5 ULN | 0 | 1 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: >10 ULN | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase: >3 ULN | 0 | 2 | 0 | 1 | 0 | 0
  Alanine Aminotransferase: >5 ULN | 0 | 1 | 0 | 0 | 0 | 0
  Alanine Aminotransferase: >10 ULN | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase > 3 ULN and Bilirubin > 2 ULN | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: >1.5 ULN | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin: >1.5 ULN | 1 | 0 | 1 | 0 | 0 | 2
  Total Bilirubin: >2 ULN | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin > 35% Bilirubin and Bilirubin > 1.5 ULN | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities in Hematology
Description: Blood samples were collected to determine the hematology laboratory significant abnormalities.
Time Frame: From first dose of IMP up to 4 weeks after the last treatment administration of the IMP, a maximum up to 458 weeks
Population: The safety analysis set included all participants who received at least 1 complete infusion of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
Participants
  Hemoglobin: <=115 g/L (Male); <=95 g/L (Female) | 1 | 0 | 1 | 0 | 0 | 1
  Hemoglobin: >=185 g/L (Male); >=165 g/L (Female) | 0 | 0 | 0 | 0 | 1 | 0
  Hemoglobin: Decrease from baseline >=20 g/L | 1 | 1 | 1 | 2 | 0 | 1
  Hematocrit: <=0.37 volume per volume (v/v) (Male); <=0.32 v/v (Female) | 1 | 0 | 1 | 1 | 1 | 1
  Hematocrit: >=0.55 v/v (Male); >=0.5 v/v (Female) | 0 | 0 | 0 | 0 | 1 | 0
  Platelet Count: <100x10^9/L | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count: >=700x10^9/L | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocyte Count: >=6x10^12/L | 0 | 0 | 0 | 0 | 1 | 0
  Monocytes: >0.7x10^9/L | 1 | 0 | 1 | 1 | 0 | 0
  Basophils: >0.1x10^9/L | 1 | 0 | 2 | 1 | 0 | 0
  Leukocyte Count: <3x10^9/L (Non-Black); <2x10^9/L (Black) | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte Count: >=16x10^9/L | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils: <1.5x10^9/L (Non-Black); <1x10^9/L (Black) | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: >4x10^9/L | 0 | 1 | 0 | 0 | 0 | 0
  Eosinophils: >0.5x10^9/L or >ULN (if ULN >=0.5x10^9/L) | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Change From Baseline in Urine BUN up to Last IMP Administration
Description: Last on-treatment (LOT) values were collected at or just prior to the last IMP administration.
Time Frame: Baseline (Day 1) and last on-treatment values (up to 454 weeks)
Population: The safety analysis set included all participants who received at least 1 complete infusion of IMP.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
millimoles per liter (mmol/L) | 60.8 (121.0) | -17.6 (268.8) | 179.5 (157.7) | 72.9 (25.8) | 37.1 (186.5) | 118.8 (134.8)

6. Primary Outcome: Change From Baseline in Urine Hyaline Casts up to Last IMP Administration
Description: The LOT values were collected at or just prior to the last IMP administration.
Time Frame: Baseline (Day 1) and last on-treatment values (up to 454 weeks)
Population: The safety analysis set included all participants who received at least 1 complete infusion of IMP. Only participants with data collected for LOT value are reported.
Measure: Mean (Standard Deviation); unit: casts per low-power field (casts/lpf)
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
casts per low-power field (casts/lpf) |  | 2.0 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  |

7. Primary Outcome: Change From Baseline in Urine Leukocytes [White Blood Cell (WBC)] up to Last IMP Administration
Description: The LOT values were collected at or just prior to the last IMP administration.
Time Frame: Baseline (Day 1) and last on-treatment values (up to 454 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: WBC per high power field (WBC/HPF)
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
WBC per high power field (WBC/HPF) |  | -1.0 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  |

8. Primary Outcome: Change From Baseline in Urine Specific Gravity up to Last IMP Administration
Description: The LOT values were collected at or just prior to the last IMP administration.
Time Frame: Baseline (Day 1) and last on-treatment values (up to 454 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
ratio | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.1) | 0.0 (0.0) | 0.0 (0.0)

9. Primary Outcome: Change From Baseline in Urine pH up to Last IMP Administration
Description: The LOT values were collected at or just prior to the last IMP administration.
Time Frame: Baseline (Day 1) and last on-treatment values (up to 454 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pH score
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 3
pH score | -0.4 (1.3) | 0.2 (1.0) | -0.3 (1.1) | 0.1 (0.5) | -0.8 (0.4) | -0.3 (0.9)

10. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Abnormalities
Description: Participants vital signs were examined to determine the abnormalities. Vital signs included heart rate, systolic and diastolic blood pressure.
Time Frame: From first dose of IMP up to 4 weeks after the last treatment administration of the IMP, a maximum up to 458 weeks
Population: The safety analysis set included all participants who received at least 1 complete infusion of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
Participants
  Systolic Blood Pressure: <=95 millimeter of mercury (mmHg) and decrease from baseline >=20 mmHg | 2 | 2 | 2 | 2 | 3 | 2
  Systolic Blood Pressure: >=160 mmHg and increase from baseline >=20 mmHg | 2 | 0 | 1 | 2 | 0 | 3
  Diastolic Blood Pressure: <=45 mmHg and decrease from baseline >=10 mmHg | 2 | 0 | 0 | 2 | 0 | 2
  Diastolic Blood Pressure: >=110 mmHg and increase from baseline >=10 mmHg | 2 | 0 | 0 | 0 | 0 | 2
  Heart Rate (HR): <=50 beats/minute (bpm) and decrease from baseline >=20 bpm | 1 | 0 | 1 | 0 | 1 | 0
  HR: >=120 bpm and increase from baseline >=20 bpm | 2 | 1 | 2 | 2 | 2 | 4

11. Primary Outcome: Number of Participants With Body Weight Increased/Decreased
Description: Body weight was measured in kilograms and collected in the electronic case report forms every 3 months throughout the duration of the study, as well as at the end of study visit.
Time Frame: From first dose of IMP up to 4 weeks after the last treatment administration of the IMP, a maximum up to 458 weeks
Population: The safety analysis set included all participants who received at least 1 complete infusion of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
Participants | 1 | 0 | 0 | 1 | 0 | 2

12. Primary Outcome: Number of Participants With Potentially Clinically Significant 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Standard 12-lead ECGs were recorded after at least 15 minutes in the supine position using an electrocardiographic device. The following were assessed: heart rate, rhythm, interval between the peaks of successive QRS complexes (RR), interval from the beginning of the P wave until the beginning of the QRS complex (PR), interval from start of the Q wave to the end of the S wave (QRS), interval between the start of the Q wave and the end of the T wave (QT), QT interval corrected for heart rate (QTc) automatic correction evaluation (by the ECG device), QRS axis, R voltage V6, voltage V1, left ventricular hypertrophy criteria, right ventricular hypertrophy criteria, repolarization charges, and overall cardiac impression for each participant.
Time Frame: From first dose of IMP up to 4 weeks after the last treatment administration of the IMP, a maximum up to 458 weeks
Population: The safety analysis set included all participants who received at least 1 complete infusion of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
Participants
  HR: <50 bpm | 1 | 0 | 0 | 0 | 1 | 0
  HR: <50 bpm and decrease from baseline >=20 bpm | 0 | 0 | 0 | 0 | 0 | 0
  HR: <40 bpm | 0 | 0 | 0 | 0 | 0 | 0
  HR: <40 bpm and decrease from baseline >=20 bpm | 0 | 0 | 0 | 0 | 0 | 0
  HR: <30 bpm | 0 | 0 | 0 | 0 | 0 | 0
  HR: <30 bpm and decrease from baseline >=20 bpm | 0 | 0 | 0 | 0 | 0 | 0
  HR: >90 bpm | 0 | 2 | 0 | 0 | 0 | 2
  HR: >90 bpm and increase from baseline >=20 bpm | 0 | 2 | 0 | 0 | 0 | 0
  HR: >100 bpm | 0 | 0 | 1 | 0 | 0 | 0
  HR: >100 bpm and increase from baseline >=20 bpm | 0 | 0 | 0 | 0 | 0 | 0
  HR: >120 bpm | 0 | 0 | 0 | 0 | 0 | 0
  HR: >120 bpm and increase from baseline >=20 bpm | 0 | 0 | 0 | 0 | 0 | 0
  PR Duration: > 200 millisecond (msec) | 0 | 1 | 1 | 0 | 0 | 1
  PR Duration: >200 msec and increase from baseline >=25% | 0 | 1 | 0 | 0 | 0 | 0
  PR Duration: >220 msec | 0 | 0 | 0 | 1 | 0 | 0
  PR Duration: >220 msec and increase from baseline >=25% | 0 | 0 | 0 | 1 | 0 | 0
  PR Duration: >240 msec | 0 | 0 | 0 | 0 | 0 | 0
  PR Duration: >240 msec and increase from baseline >=25% | 0 | 0 | 0 | 0 | 0 | 0
  QRS Duration: >110 msec | 0 | 0 | 1 | 0 | 3 | 4
  QRS Duration: >110 msec and increase from baseline >=25% | 0 | 0 | 0 | 0 | 0 | 0
  QRS Duration: >120 msec | 0 | 1 | 1 | 1 | 0 | 0
  QRS Duration: >120 msec and increase from baseline >=25% | 0 | 0 | 1 | 0 | 0 | 0
  QTcB - Bazett's Correction Formula: >450 msec | 1 | 1 | 1 | 2 | 1 | 3
  QTcB - Bazett's Correction Formula: >480 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcB - Bazett's Correction Formula: >500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcB - Bazett's Correction Formula: Increase from baseline (30-60) msec | 0 | 2 | 1 | 1 | 1 | 4
  QTcB - Bazett's Correction Formula: Increase from baseline >60 msec | 0 | 0 | 0 | 0 | 1 | 0
  QTcF - Fridericia's Correction Formula: >450 msec | 0 | 1 | 0 | 1 | 1 | 0
  QTcF - Fridericia's Correction Formula: >480 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF - Fridericia's Correction Formula: >500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF - Fridericia's Correction Formula: Increase from baseline (30-60) msec | 0 | 1 | 0 | 0 | 0 | 1
  QTcF - Fridericia's Correction Formula: Increase from baseline >60 msec | 0 | 0 | 0 | 0 | 1 | 0

13. Primary Outcome: Number of Participants With Antidrug Antibodies (ADA) Status, Positive or Negative
Description: ADA negative was defined as ADAs are not detected (that is, negative in screening assay or reactive in screening but negative in confirmatory assay). ADA positive was defined as ADA was detected (that is, an assay signal equal to or greater than the cut-point in the screening assay and was tested positive in the confirmatory assay).
Time Frame: From first dose of IMP up to 4 weeks after the last treatment administration of the IMP, a maximum up to 458 weeks
Population: The Pharmacodynamic (PD) analysis set included enrolled participants without any critical deviations related to IMP administration, and for whom any PD data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
Participants
  ADA negative | 0 | 1 | 0 | 1 | 1 | 3
  ADA positive at baseline | 0 | 0 | 0 | 1 | 3 | 1
  ADA positive post-baseline | 4 | 2 | 3 | 2 | 0 | 2

14. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Avalglucosidase Alfa
Description: Cmax was defined as maximum plasma concentration observed. The non-compartmental pharmacokinetic (PK) analysis was performed.
Time Frame: Predose (prior to infusion), end of the infusion and at 1, 4, 8, 12, and 24 hours post-dose on Week 312
Population: The PK analysis set included enrolled participants without any critical deviations related to IMP administration, and for whom any PK data were available. As pre-specified, results for this outcome measure are presented combinedly for all the dosage groups (5, 10 and 20 mg/kg) under the corresponding reporting groups, Group 1: (Avalglucosidase Alfa) and Group 2: (Avalglucosidase Alfa).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Groups:
- Group 1: Avalglucosidase Alfa: Participants who were treatment-naïve to alglucosidase alfa received avalglucosidase alfa 5 or 10 or 20 mg/kg IV infusion qow for up to 454 weeks.
- Group 2: Avalglucosidase Alfa: Participants who were previously treated with alglucosidase alfa received avalglucosidase alfa 5 or 10 or 20 mg/kg IV infusion qow for up to 450 weeks.
Arm/Group | Group 1: Avalglucosidase Alfa | Group 2: Avalglucosidase Alfa
Number analyzed (Participants) | 4 | 5
microgram per milliliter (mcg/mL) | 269 (16) | 234 (24)

15. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Real Time (AUClast) of Avalglucosidase Alfa
Description: AUClast was calculated using the trapezoidal method from time zero to the real time. The non-compartmental PK analysis was performed.
Time Frame: Predose (prior to infusion), end of the infusion and at 1, 4, 8, 12, and 24 hours post-dose on Week 312
Population: The PK analysis set included enrolled participants without any critical deviations related to IMP administration, and for whom any PK data were available. As pre-specified, results for this outcome measure are presented combinedly for all dosage groups (5, 10 and 20 mg/kg) under corresponding reporting groups, Group 1: (Avalglucosidase Alfa) and Group 2: (Avalglucosidase Alfa). Overall Number of Participants Analyzed = Number of participants contributed to the analysis for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*mcg/mL
Arm/Group | Group 1: Avalglucosidase Alfa | Group 2: Avalglucosidase Alfa
Number analyzed (Participants) | 4 | 4
hour*mcg/mL | 1350 (24) | 1290 (21)

16. Primary Outcome: Time Corresponding to the Last Concentration (Tlast) of Avalglucosidase Alfa
Description: Tlast was defined as time corresponding to the last concentration above the limit of quantification, Clast. The non-compartmental PK analysis was performed.
Time Frame: Predose (prior to infusion), end of the infusion and at 1, 4, 8, 12, and 24 hours post-dose on Week 312
Population: as for outcome 15
Measure: Median (Full Range); unit: hour
Arm/Group | Group 1: Avalglucosidase Alfa | Group 2: Avalglucosidase Alfa
Number analyzed (Participants) | 4 | 4
hour | 25.84 [25.65 to 27.73] | 27.6 [7.5 to 29.5]

17. Primary Outcome: Terminal Half-Life (t1/2z) of Avalglucosidase Alfa
Description: t1/2z was calculated according to the following equation: t1/2z = 0.693/λz. Where, λz is the slope of the regression line of the terminal phase of the plasma concentration versus time curve. Half-life was calculated by taking the regression of at least 3 points. The non-compartmental PK analysis was performed.
Time Frame: Predose (prior to infusion), end of the infusion and at 1, 4, 8, 12, and 24 hours post-dose on Week 312
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Group 1: Avalglucosidase Alfa | Group 2: Avalglucosidase Alfa
Number analyzed (Participants) | 4 | 4
hour | 1.62 (9) | 1.79 (8)

18. Primary Outcome: Apparent Total Body Clearance Steady-State (CLss) of Avalglucosidase Alfa
Description: CLss was calculated using the following equation: CLss= dose/AUC. The non-compartmental PK analysis was performed.
Time Frame: Predose (prior to infusion), end of the infusion and at 1, 4, 8, 12, and 24 hours post-dose on Week 312
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Group 1: Avalglucosidase Alfa | Group 2: Avalglucosidase Alfa
Number analyzed (Participants) | 4 | 3
liter/hour | 0.90 (24) | 1.06 (12)

19. Primary Outcome: Apparent Volume of Distribution Steady-State (Vss) of Avalglucosidase Alfa
Description: Vss was calculated using the following equation: Vz= CLss/λz. The non-compartmental PK analysis was performed.
Time Frame: Predose (prior to infusion), end of the infusion and at 1, 4, 8, 12, and 24 hours post-dose on Week 312
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Group 1: Avalglucosidase Alfa | Group 2: Avalglucosidase Alfa
Number analyzed (Participants) | 4 | 3
liter | 3.04 (13) | 3.8 (24)

20. Secondary Outcome: Change From Baseline in Cross-Sectional Area (CSA) of Skeletal Muscle Magnetic Resonance Imaging (MRI) Up to Week 442
Description: Skeletal muscle MRI performed prior to the muscle needle or open biopsy procedure using both qualitative (T1) and quantitative (T2, dixon) modalities to assess disease severity and detect treatment effects. The T1 weighted axial data was analyzed using the mercuri scale, which determines degree of intact muscle and fatty replacement, providing a qualitative measure of overall disease severity. Trophicity changes were evaluated for 5 muscle groups, including the upper leg muscles (quadriceps, hamstring) and the lower leg muscles (triceps, extensors, fibularis). The measured area of each muscle group, CSA was provided.
Time Frame: Baseline (Day 1) and Weeks 104 and 442
Population: The PD analysis set included enrolled participants without any critical deviations related to IMP administration, and for whom any PD data were available. Only participants with data collected at specific time points are reported.
Measure: Mean (Standard Deviation); unit: millimeter square (mm^2)
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 2 | 3
millimeter square (mm^2)
  Week 104: CSA - Fibularis muscle |  |  | 57.4 (3.9) | -0.9 (46.9) | 46.1 (81.2) | 26.7 (40.0)
  Week 104: CSA - Hamstring muscle |  |  | 123.0 (254.7) | -135.7 (138.7) | 70.6 (368.1) | 215.2 (126.1)
  Week 104: CSA - Leg extensor muscle |  |  | 23.2 (60.2) | 23.1 (19.1) | 107.9 (145.0) | 39.1 (26.6)
  Week 104: CSA - Quadriceps muscle |  |  | 303.3 (49.5) | -27.6 (45.8) | 134.0 (569.4) | 193.3 (103.3)
  Week 104: CSA - Triceps surae muscle |  |  | 283.6 (123.7) | -310.0 (383.2) | -3.5 (334.6) | 226.0 (172.3)
  Week 442: CSA - Fibularis muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: CSA - Fibularis muscle |  |  |  |  | -41.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -55.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: CSA - Hamstring muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: CSA - Hamstring muscle |  |  |  |  | -461.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -30.2 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: CSA - Leg extensor muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: CSA - Leg extensor muscle |  |  |  |  | -102.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -68.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: CSA - Quadriceps muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: CSA - Quadriceps muscle |  |  |  |  | -644.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 19.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: CSA - Triceps surae muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: CSA - Triceps surae muscle |  |  |  |  | -220.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -82.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.

21. Secondary Outcome: Change From Baseline in Dixon Fat Fraction of Skeletal Muscle Magnetic Resonance Imaging (MRI) Up to Week 442
Description: Skeletal muscle MRI performed prior to the muscle needle or open biopsy procedure using both qualitative (T1) and quantitative (T2, dixon) modalities to assess disease severity and detect treatment effects. The T1 weighted axial data was analyzed using the mercuri scale, which determines degree of intact muscle and fatty replacement, providing a qualitative measure of overall disease severity. Trophicity changes were evaluated for 5 muscle groups, including the upper leg muscles (quadriceps, hamstring) and the lower leg muscles (triceps, extensors, fibularis). Three-point dixon imaging provided quantification of fat content in muscles [fat fraction (FF)].
Time Frame: Baseline (Day 1) and Weeks 104 and 442
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 3
percentage (%)
  Week 104: Dixon fat fraction - Fibularis muscle |  |  | 0.9 (0.1) | 1.4 (2.2) | -0.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.3 (1.1)
  Week 104: Dixon fat fraction - Hamstring muscle |  |  | 5.7 (3.3) | -0.2 (2.6) | -0.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 3.4 (3.9)
  Week 104: Dixon fat fraction - Leg extensor muscle |  |  | 0.9 (0.1) | 0.8 (2.2) | -0.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -0.2 (1.3)
  Week 104: Dixon fat fraction - Quadriceps muscle |  |  | 2.3 (1.4) | -0.5 (2.3) | 0.2 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 2.4 (3.6)
  Week 104: Dixon fat fraction - Triceps surae muscle |  |  | 0.4 (0.3) | 1.4 (1.7) | -0.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.9 (0.5)
  Week 442: Dixon fat fraction - Fibularis muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: Dixon fat fraction - Fibularis muscle |  |  |  |  | 2.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: Dixon fat fraction - Hamstring muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: Dixon fat fraction - Hamstring muscle |  |  |  |  | 10.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: Dixon fat fraction - Leg extensor muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: Dixon fat fraction - Leg extensor muscle |  |  |  |  | 1.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -0.0 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: Dixon fat fraction - Quadriceps muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: Dixon fat fraction - Quadriceps muscle |  |  |  |  | 9.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: Dixon fat fraction - Triceps surae muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: Dixon fat fraction - Triceps surae muscle |  |  |  |  | 1.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.

22. Secondary Outcome: Change From Baseline in Index of Real Muscle Mass (IRMM) of Skeletal Muscle Magnetic Resonance Imaging (MRI) Up to Week 442
Description: Skeletal muscle MRI performed prior to the muscle needle or open biopsy procedure using both qualitative (T1) and quantitative (T2, dixon) modalities to assess disease severity and detect treatment effects. The T1 weighted axial data was analyzed using the mercuri scale, which determines degree of intact muscle and fatty replacement, providing a qualitative measure of overall disease severity. Trophicity changes were evaluated for 5 muscle groups, including the upper leg muscles (quadriceps, hamstring) and the lower leg muscles (triceps, extensors, fibularis). The FF was combined with the CSA measurements trophicity to provide an IRMM in mm^2 (that is, IRMM = CSA x [1 - FF]). A negative change from baseline value in IRMM of skeletal muscle MRI indicates muscle loss (worse outcome) and a positive change from baseline value indicates muscle gain (better outcome).
Time Frame: Baseline (Day 1) and Weeks 104 and 442
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 3
mm^2
  Week 104: IRMM - Fibularis muscle |  |  | 44.8 (8.3) | -13.8 (40.4) | -5.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 21.8 (41.6)
  Week 104: IRMM - Hamstring muscle |  |  | -131.6 (77.0) | -100.9 (150.3) | -149.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 49.2 (139.0)
  Week 104: IRMM - Leg extensor muscle |  |  | 12.4 (59.9) | 9.8 (34.2) | 7.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 34.9 (33.2)
  Week 104: IRMM - Quadriceps muscle |  |  | 149.2 (135.2) | -9.4 (65.9) | -256.0 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 120.7 (166.3)
  Week 104: IRMM - Triceps surae muscle |  |  | 236.8 (122.2) | -299.6 (402.6) | -210.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 181.4 (143.7)
  Week 442: IRMM - Fibularis muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: IRMM - Fibularis muscle |  |  |  |  | -53.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -54.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: IRMM - Hamstring muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: IRMM - Hamstring muscle |  |  |  |  | -412.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -44.0 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: IRMM - Leg extensor muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: IRMM - Leg extensor muscle |  |  |  |  | -109.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -64.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: IRMM - Quadriceps muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: IRMM - Quadriceps muscle |  |  |  |  | -1085.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -21.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: IRMM - Triceps surae muscle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Week 442: IRMM - Triceps surae muscle |  |  |  |  | -288.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -85.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.

23. Secondary Outcome: Change From Baseline in T2 of Skeletal Muscle Magnetic Resonance Imaging (MRI) Up to Week 442
Description: Skeletal muscle MRI performed prior to the muscle needle or open biopsy procedure using both qualitative (T1) and quantitative (T2, dixon) modalities to assess disease severity and detect treatment effects. The T1 weighted axial data was analyzed using the mercuri scale, which determines degree of intact muscle and fatty replacement, providing a qualitative measure of overall disease severity. Trophicity changes were evaluated for 5 muscle groups, including the upper leg muscles (quadriceps, hamstring) and the lower leg muscles (triceps, extensors, fibularis). The T2 multi-slice multi-spin echo and B1 mapping provided a quantitative measure of disease activity (edema, inflammation) within muscles.
Time Frame: Baseline (Day 1) and Weeks 104 and 442
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 1 | 0 | 2 | 3 | 1 | 3
milliseconds (ms)
  Week 104: T2 - Fibularis muscle: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 3
  Week 104: T2 - Fibularis muscle |  |  | -0.6 (0.6) | 0.5 (2.4) | 0.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.0 (0.6)
  Week 104: T2 - Hamstring muscle: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1 | 3
  Week 104: T2 - Hamstring muscle |  |  | 0.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 1.6 (3.2) | -1.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.2 (0.7)
  Week 104: T2 - Leg extensor muscle: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 3
  Week 104: T2 - Leg extensor muscle |  |  | -0.8 (1.6) | 2.0 (2.2) | 1.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -0.3 (0.7)
  Week 104: T2 - Quadriceps muscle: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 3
  Week 104: T2 - Quadriceps muscle |  |  | 0.8 (1.0) | 0.5 (2.7) | -1.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 1.0 (0.6)
  Week 104: T2 - Triceps surae muscle: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 3
  Week 104: T2 - Triceps surae muscle |  |  | -0.3 (0.3) | 0.5 (1.7) | -0.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.4 (0.6)
  Week 442: T2 - Fibularis muscle: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 1
  Week 442: T2 - Fibularis muscle | -4.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  | 0.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: T2 - Hamstring muscle: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 1
  Week 442: T2 - Hamstring muscle | -6.0 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  | -9.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 2.2 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: T2 - Leg extensor muscle: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 1
  Week 442: T2 - Leg extensor muscle | -2.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  | 1.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: T2 - Quadriceps muscle: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 1
  Week 442: T2 - Quadriceps muscle | -0.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  | 1.0 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 3.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: T2 - Triceps surae muscle: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 1
  Week 442: T2 - Triceps surae muscle | -3.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  | 1.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -0.0 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.

24. Secondary Outcome: Change From Baseline in T2 With B1 of Skeletal Muscle Magnetic Resonance Imaging (MRI) Up to Week 442
Description: as for outcome 23
Time Frame: Baseline (Day 1) and Weeks 104 and 442
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 1 | 0 | 2 | 3 | 1 | 2
milliseconds (ms)
  Week 104: T2 with B1 - Fibularis muscle: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 1
  Week 104: T2 with B1 - Fibularis muscle |  |  | -0.5 (0.7) | 0.5 (2.2) | 1.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 104: T2 with B1 - Hamstring muscle: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1 | 2
  Week 104: T2 with B1 - Hamstring muscle |  |  | -0.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 2.3 (4.6) | -2.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -0.4 (1.6)
  Week 104: T2 with B1 - Leg extensor muscle: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 1
  Week 104: T2 with B1 - Leg extensor muscle |  |  | -0.6 (1.9) | 2.0 (2.2) | 0.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -2.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 104: T2 with B1 - Quadriceps muscle: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 2
  Week 104: T2 with B1 - Quadriceps muscle |  |  | 0.9 (0.7) | 0.7 (2.8) | -1.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 1.6 (0.6)
  Week 104: T2 with B1 - Triceps surae muscle: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1 | 1
  Week 104: T2 with B1 - Triceps surae muscle |  |  | -0.3 (0.4) | 0.1 (1.2) | -1.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | 0.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: T2 with B1 - Fibularis muscle: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 442: T2 with B1 - Fibularis muscle | -4.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  |  |
  Week 442: T2 with B1 - Leg extensor muscle: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 442: T2 with B1 - Leg extensor muscle | -3.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  |  |
  Week 442: T2 with B1 - Quadriceps muscle: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 442: T2 with B1 - Quadriceps muscle | -0.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  |  |
  Week 442: T2 with B1 - Triceps surae muscle: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 442: T2 with B1 - Triceps surae muscle | -3.2 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  |  |

25. Secondary Outcome: Change From Baseline in Skeletal Muscle Biopsy Up to Week 312
Description: Skeletal muscle needle or open biopsy was performed on the lower extremity (quadriceps) muscle to assess glycogen content. The MRI appearance of the muscle was used to determine the level (axial slice position) that the biopsy procedure should target (avoiding fatty replaced tissue). Glycogen content was measured by histomorphometric analysis or severity grading to determine how effectively avalglucosidase alfa was able to remove glycogen from muscle.
Time Frame: Baseline (Day 1) and Weeks 27, 104, 208, 260 and 312
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percentage of glycogen
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
percentage of glycogen
  Left quadriceps muscle: Week 27: number analyzed (Participants) | 1 | 0 | 2 | 3 | 1 | 3
  Left quadriceps muscle: Week 27 | 0.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  | 0.9 (0.1) | -3.6 (6.4) | 0.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -0.4 (0.4)
  Left quadriceps muscle: Week 104: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0
  Left quadriceps muscle: Week 104 |  |  |  | -4.8 (9.9) |  |
  Left quadriceps muscle: Week 260: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Left quadriceps muscle: Week 260 |  |  |  | -4.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |
  Right quadriceps muscle: Week 27: number analyzed (Participants) | 3 | 2 | 1 | 0 | 2 | 0
  Right quadriceps muscle: Week 27 | -1.7 (3.3) | 0.5 (1.5) | -1.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  | 2.0 (1.0) |
  Right quadriceps muscle: Week 104: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Right quadriceps muscle: Week 104 |  |  |  |  | -2.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |
  Right quadriceps muscle: Week 208: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Right quadriceps muscle: Week 208 |  |  |  |  | -3.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |
  Right quadriceps muscle: Week 312: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Right quadriceps muscle: Week 312 |  |  |  |  | -5.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |

26. Secondary Outcome: Change From Baseline in Urinary Glucose Tetrasaccharide (Hex4) Level Up to Week 442
Description: The Hex4, a tetraglucose oligomer, has been shown to be elevated in the urine of participants with Pompe disease. Hence, determination of Hex4 levels may be a means by which the efficacy of treatments were monitored. Urine samples were collected prior to IMP infusion for the assessment of urinary Hex4 concentrations.
Time Frame: Baseline (Day 1) and Weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 52, 78, 104, 130, 156, 182, 208, 234, 260, 286, 312, 338, 364, 390, 416 and 442
Population: The PD analysis set included enrolled participants without any critical deviations related to IMP administration, and for whom any PD data were available.
Measure: Mean (Standard Deviation); unit: mmol per mole
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 6
mmol per mole
  Week 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 1 | 0.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  |  |
  Week 3: number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 6
  Week 3 | -0.6 (0.2) | -1.9 (1.6) | -0.9 (0.5) | -0.9 (1.0) | -0.5 (1.1) | -0.2 (1.5)
  Week 5: number analyzed (Participants) | 4 | 3 | 3 | 4 | 4 | 5
  Week 5 | -1.0 (0.5) | -0.2 (0.4) | -1.0 (1.1) | 0.2 (0.7) | -0.5 (1.1) | -1.5 (2.0)
  Week 7 | -1.2 (1.1) | -2.2 (1.7) | -0.6 (1.3) | -0.7 (0.8) | -0.3 (1.1) | -1.2 (2.3)
  Week 9 | -0.6 (1.7) | -2.4 (3.2) | 0.5 (0.7) | 0.0 (1.3) | -0.7 (1.3) | -2.2 (2.7)
  Week 11 | -0.1 (1.9) | -2.7 (2.6) | 0.4 (1.0) | 0.1 (0.8) | -0.5 (1.7) | -2.5 (3.3)
  Week 13 | -1.3 (1.3) | -5.0 (3.4) | -1.6 (1.5) | 0.5 (0.7) | -0.7 (1.3) | -2.7 (3.6)
  Week 15 | -1.4 (0.5) | -6.2 (3.3) | -1.4 (0.5) | 0.6 (1.5) | -1.0 (1.3) | -3.4 (4.8)
  Week 17: number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 5
  Week 17 | -1.0 (0.3) | -6.7 (2.1) | -1.5 (1.2) | -0.0 (1.4) | -0.9 (1.3) | -3.4 (4.5)
  Week 19: number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 5
  Week 19 | -2.3 (2.4) | -6.5 (2.5) | -1.6 (1.0) | 0.3 (3.1) | -0.8 (1.8) | -4.0 (5.9)
  Week 21: number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 5
  Week 21 | -2.3 (2.1) | -6.5 (2.2) | -1.8 (1.3) | 0.1 (2.2) | -0.8 (1.7) | -4.4 (5.6)
  Week 23: number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 5
  Week 23 | -1.7 (1.7) | -5.3 (1.3) | -0.7 (1.4) | 0.7 (3.1) | -0.9 (1.9) | -2.9 (5.5)
  Week 25: number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 5
  Week 25 | -2.5 (3.0) | -4.5 (1.0) | -1.3 (2.3) | 0.3 (3.7) | -0.8 (1.9) | -3.1 (5.0)
  Week 27: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 27 | -2.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  |  |
  Week 52: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 5
  Week 52 | -1.8 (1.6) | -4.1 (5.2) | -2.0 (2.0) | 0.2 (2.7) | -1.2 (2.0) | -3.4 (5.4)
  Week 78: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 5
  Week 78 | -1.9 (1.3) | -3.5 (5.0) | -2.9 (3.2) | -0.9 (2.4) | -1.5 (1.8) | -3.5 (5.5)
  Week 104: number analyzed (Participants) | 3 | 1 | 3 | 3 | 3 | 5
  Week 104 | -3.0 (2.9) | -6.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -2.8 (3.4) | 0.8 (3.8) | -1.9 (1.5) | -3.6 (4.1)
  Week 130: number analyzed (Participants) | 3 | 1 | 3 | 2 | 3 | 5
  Week 130 | -4.0 (3.9) | -9.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -2.4 (3.3) | -1.4 (3.9) | -1.9 (1.6) | -3.1 (3.9)
  Week 156: number analyzed (Participants) | 3 | 1 | 3 | 3 | 3 | 4
  Week 156 | -3.6 (3.1) | -10.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -1.9 (3.2) | -1.4 (3.2) | -2.6 (1.8) | -4.8 (7.9)
  Week 182: number analyzed (Participants) | 3 | 1 | 3 | 3 | 2 | 5
  Week 182 | -3.5 (2.6) | -11.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -2.2 (2.7) | -3.1 (3.2) | -1.8 (0.4) | -3.9 (6.5)
  Week 208: number analyzed (Participants) | 3 | 1 | 3 | 3 | 3 | 4
  Week 208 | -3.2 (3.2) | -6.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -2.6 (3.9) | -3.9 (3.5) | -1.7 (0.6) | -5.9 (9.5)
  Week 234: number analyzed (Participants) | 3 | 1 | 1 | 3 | 3 | 4
  Week 234 | -3.4 (3.2) | -3.8 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -4.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -4.1 (2.5) | -2.9 (1.2) | -4.9 (7.1)
  Week 260: number analyzed (Participants) | 2 | 1 | 3 | 2 | 3 | 4
  Week 260 | -1.9 (0.4) | -10.1 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -1.7 (4.0) | -5.9 (0.1) | -2.9 (1.7) | -5.6 (8.8)
  Week 286: number analyzed (Participants) | 1 | 0 | 0 | 2 | 2 | 1
  Week 286 | -7.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  | -3.6 (2.2) | -2.0 (0.6) | -0.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 312: number analyzed (Participants) | 3 | 0 | 2 | 2 | 2 | 2
  Week 312 | -3.6 (3.0) |  | -4.3 (3.9) | -4.6 (1.9) | -1.9 (0.7) | -2.0 (0.2)
  Week 338: number analyzed (Participants) | 0 | 1 | 2 | 1 | 2 | 4
  Week 338 |  | -0.4 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -4.2 (5.5) | -4.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -1.8 (0.4) | -5.7 (8.2)
  Week 364: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 364 | -2.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  |  |
  Week 390: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 2
  Week 390 | -2.6 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  | -1.3 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  | -10.5 (11.7)
  Week 416: number analyzed (Participants) | 0 | 1 | 2 | 2 | 1 | 1
  Week 416 |  | -12.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -1.9 (3.2) | -4.7 (2.5) | -2.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -0.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.
  Week 442: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 1
  Week 442 | -8.5 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. |  |  |  | -1.9 (NA) — Standard deviation could not be determined when only 1 participant is analyzed. | -0.7 (NA) — Standard deviation could not be determined when only 1 participant is analyzed.

ADVERSE EVENTS:
Time Frame: TEAEs data was collected from first dose of IMP up to 4 weeks after the last dose of IMP administration (maximum exposure duration: up to 454 weeks). Death data were collected from first dose of IMP up to the end of the study.
Description: Analysis was performed on the safety analysis set.
Arm/Group | Group 1: Avalglucosidase Alfa 5 mg/kg | Group 1: Avalglucosidase Alfa 10 mg/kg | Group 1: Avalglucosidase Alfa 20 mg/kg | Group 2: Avalglucosidase Alfa 5 mg/kg | Group 2: Avalglucosidase Alfa 10 mg/kg | Group 2: Avalglucosidase Alfa 20 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 1/3 | 0/4 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/3 | 1/3 | 1/4 | 1/4 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 4/4 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Avalglucosidase Alfa 5 mg/kg (N=4) | Group 1: Avalglucosidase Alfa 10 mg/kg (N=3) | Group 1: Avalglucosidase Alfa 20 mg/kg (N=3) | Group 2: Avalglucosidase Alfa 5 mg/kg (N=4) | Group 2: Avalglucosidase Alfa 10 mg/kg (N=4) | Group 2: Avalglucosidase Alfa 20 mg/kg (N=6)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fractured Sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postimplantation Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram Q Wave Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labour Pain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic Dilatation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extravasation Blood (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral Artery Stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Avalglucosidase Alfa 5 mg/kg (N=4) | Group 1: Avalglucosidase Alfa 10 mg/kg (N=3) | Group 1: Avalglucosidase Alfa 20 mg/kg (N=3) | Group 2: Avalglucosidase Alfa 5 mg/kg (N=4) | Group 2: Avalglucosidase Alfa 10 mg/kg (N=4) | Group 2: Avalglucosidase Alfa 20 mg/kg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conduction Disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral Valve Prolapse (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia Paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness Unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid Ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling Of Eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 2 (5) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (10) | 1 (3) | 3 (3) | 2 (4) | 1 (3) | 2 (2)
Diverticulum Intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip Haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malpositioned Teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (13) | 1 (1) | 1 (1) | 2 (4) | 1 (2) | 1 (2)
Oral Mucosal Blistering (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic Ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swollen Tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application Site Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (8)
Catheter Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (5) | 2 (4) | 0 (0) | 1 (3) | 0 (0) | 3 (6)
Feeling Hot (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired Healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Infusion Site Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion Site Rash (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion Site Swelling (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection Site Haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection Site Swelling (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (2)
Peripheral Swelling (General disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (9) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Vaccination Site Reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Fibrosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy To Arthropod Bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Ear Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Eye Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (6) | 2 (6) | 2 (8) | 4 (8) | 3 (5) | 2 (10)
Oral Herpes (Infections and infestations) | 2 (14) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 2 (3)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (4) | 0 (0) | 1 (1) | 1 (4) | 1 (1) | 3 (8)
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adverse Event Following Immunisation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avulsion Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Electric Shock (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 3 (8) | 0 (0) | 1 (1) | 4 (11) | 1 (1) | 4 (19)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iliotibial Band Syndrome (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Antimitochondrial Antibody Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Antinuclear Antibody Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Calcium Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Chloride Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood Lactic Acid Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Potassium Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Potassium Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Sodium Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Urea Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body Temperature Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath Sounds Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular Pressure Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoprotein (A) Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pulmonary Function Test Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcus Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin T Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine Analysis Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (8) | 1 (1) | 1 (2) | 3 (5) | 1 (1) | 4 (21)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 3 (10)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diffuse Idiopathic Skeletal Hyperostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Greater Trochanteric Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaw Clicking (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 (8) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (11) | 1 (15) | 1 (3) | 2 (9) | 0 (0) | 3 (6)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (9)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cervical Radiculopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (12) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 2 (4)
Dizziness Postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (15) | 2 (12) | 2 (8) | 2 (16) | 0 (0) | 2 (22)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Migraine With Aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sedation Complication (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory Loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tension Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Afterbirth Pain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device Occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Delusional Disorder, Persecutory Type (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine Flow Decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Endometrial Thickening (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic Respiratory Symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3) | 0 (0) | 1 (1) | 1 (2) | 1 (3)
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restrictive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal Polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myxoid Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (9) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pregnancy Of Partner (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (7)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (9) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-11-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT02032524/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT02032524/SAP_001.pdf